CLINICAL TRIAL: NCT03698669
Title: Treating Chronic Pain in Buprenorphine Patients in Primary Care Settings
Acronym: TOPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-38056; 1R01DA045695 (NIH)
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Opioid-Related Disorders
Keywords: Depression; Pain; Cognitive behavioral therapy (CBT); Buprenorphine; Behavioral health specialist (BHS); Primary care provider (PCP)
MeSH Terms: conditions — Opioid-Related Disorders; Depression; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treating Opioid Patients' Pain and Sadness (TOPPS) (Experimental): TOPPS, consists of three main components: (1) psychoeducation about pain, depression, opioid use, their interactions, and the maintaining role of avoidance; (2) coaching in being an informed, activated patient (based in part on the chronic care model and on approaches to self-management of chronic illness); and (3) behavioral activation to increase engagement in meaningful activities.
  Interventions: Behavioral: Treating Opioid Patients' Pain and Sadness (TOPPS)
- Health Education (HE) (Active Comparator): Participants randomized to the control HE condition are offered six telephone sessions led by the Behavioral Health Specialists. The first health session is around nutrition. At the remaining sessions, participants choose from a menu of topics, including: a second session on nutrition; germs, colds and the flu; preventing cancer; diabetes; protecting your heart; getting a good night's sleep; complementary and alternative medicine; caffeine, or physical activity.
  Interventions: Behavioral: Health Education (HE)

INTERVENTIONS:
Behavioral: Treating Opioid Patients' Pain and Sadness (TOPPS) — TOPPS, consists of three main components: (1) psychoeducation about pain, depression, opioid use, their interactions, and the maintaining role of avoidance; (2) coaching in being an informed, activated patient (based in part on the chronic care model and on approaches to self-management of chronic illness); and (3) behavioral activation to increase engagement in meaningful activities.
  Arms: Treating Opioid Patients' Pain and Sadness (TOPPS)
Behavioral: Health Education (HE) — Participants randomized to the control HE condition are offered six telephone sessions led by the Behavioral Health Specialists. The first health session is around nutrition. At the remaining sessions, participants choose from a menu of topics, including: a second session on nutrition; germs, colds and the flu; preventing cancer; diabetes; protecting your heart; getting a good night's sleep; complementary and alternative medicine; caffeine, or physical activity.
  Arms: Health Education (HE)

SUMMARY:
Treating Opioid Patients' Pain and Sadness (TOPPS) focuses on the relationship of pain, depression, opioid and other substance misuse, and functioning. It has a structured agenda, uses behavioral activation, involves explicit and ongoing psychoeducation, and includes a behavioral health specialist (BHS) trained extensively in the nature of pain and opioid misuse, including how to assess for red flags of opioid relapse. Devised specifically for primary care patients receiving buprenorphine, TOPPS is collaborative (PCP, BHS, and patient) and focuses on pain and physical symptoms in order to decrease the need to turn to substance misuse to avoid pain, and to foster patient's abilities to achieve their long-term life goals. In this study, TOPPS is compared to a health education contact-control condition among 250 persons with opioid use disorder recruited from two primary care based buprenorphine programs. The investigators will provide both interventions over 3 months, and follow the patients for a total of 12 months in order to observe both short-term and longer-term effects of TOPPS.

DETAILED DESCRIPTION:
Nearly 2.5 million individuals in the United States have opioid use disorder (OUD), with the vast majority (2 million) reporting abuse of prescription opioids. Patients with a history of substance use are particularly vulnerable to experiencing pain. Indeed, a large percentage of patients with OUD who receive the effective opioid agonist treatments (OAT) buprenorphine or methadone (MMT), report that pain preceded any use of addictive substances, and that the primary reason for starting opioid use was to reduce pain. Among methadone patients, 37-61% suffer from chronic pain that is often severe and interferes with daily activities. Similarly, in studies of chronic pain in buprenorphine patients, approximately 48% of patients report chronic pain. OAT recipients report far higher rates of chronic pain than the wider US population.

Chronic pain has been associated with negative substance use outcomes in persons receiving buprenorphine for opioid detoxification and in people receiving MMT. Providers may prioritize the treatment of substance use in OUD patients, leaving the concurrent pain untreated. Lack of treatment encourages patients to use illicit opioids for pain relief. Indeed, for persons using buprenorphine, greater pain severity in a given week was significantly associated with increased likelihood of opioid use in the following week.

Pain contributes to other negative outcomes. Pain is an independent risk factor for suicide including in samples of substance use disorder patients. Further, compared to MMT patients without pain, those with pain have significantly greater health problems and psychological distress. Pain, poor health, and low energy are the most commonly cited reasons that OAT patients are physically inactive. The continued physical and social problems in patients with pain influence the perception of (lack of) treatment benefits by both patients and providers.

Duration of opioid agonist treatment (OAT) is a key predictor of long-term abstinence and outcomes improve across a variety of domains if patients remain in care for at least one year. Although buprenorphine is a growing ambulatory treatment, retention in care remains problematic. Across practice sites and, despite variations in visit frequency, the 12-month retention rate ranges from 50-80% with the majority of treatment drop-out occurring during the first three months of treatment. Though few studies have yet examined the role of pain, pain has been found to negatively impact buprenorphine treatment retention.

Studies estimate that approximately one third to one half of MMT and buprenorphine recipients suffer from depression. Several studies have reported that opioid dependent patients with chronic pain have greater depressive symptoms and a greater probability of occupational disability compared to patients with lower level or no chronic pain. Amongst MMT patients, higher psychiatric distress is associated with lower general functioning. Methadone counselors report difficulty treating patients with chronic pain due in part to these patients' co-occurring psychiatric symptoms. In the only study of antidepressant treatment for depressed persons initiating buprenorphine, the investigators found in a secondary analysis that pain is prevalent, interferes with functioning, and its severity plateaus after one month of buprenorphine. Importantly, as with chronic pain, depressive symptoms have been associated with greater likelihood of relapse to opioid use in OAT patients. The substantial overlap of pain and depression in OAT patients suggest that functioning may improve most when depression and pain are simultaneously treated in an integrated fashion that is theoretically-based.

TOPPS is a type of cognitive behavioral therapy (CBT) that consists of three main components: 1) psychoeducation about pain, depression, opioid misuse, their interaction, and the maintaining role of avoidance; 2) coaching in being an informed, activated patient; and 3) behavioral activation with a focus on acceptance. Modern behavioral activation is idiographic and responsive to each patient's unique environment, needs, and goals. The function of a behavior is analyzed, and if the function is avoidance (e.g., of social contact, personal engagement, or physical activity), the behavior is targeted for change. Patients are taught to consider behavioral options, and to choose an option inconsistent with avoidance. There is an implicit attitude of acceptance of thoughts and feelings, as behavior is not dependent on changing thoughts and feelings. Behavior activation for depression focuses on helping patients to set goals in meaningful life areas, and then to break down long-term goals into smaller weekly goals. This process is incompatible with behavioral avoidance and instead, encourages patients to approach meaningful life goals. Barriers that arise in achieving short-term goals are addressed in treatment.

TOPPS focuses on the relationship of pain, depression, opioid and other substance misuse, and functioning. It has a structured agenda, uses behavioral activation, involves explicit and ongoing psychoeducation, and includes a BHS trained extensively in the nature of pain and opioid misuse and relapse. Devised specifically for primary care patients receiving buprenorphine, TOPPS is collaborative (physician, interventionist, and patient) and focuses on depression, pain and physical symptoms in order to decrease the need to turn to substance misuse to avoid pain, increase overall functioning and to foster patient's abilities to achieve their long-term life goals.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 65 years of age
2. Have chronic pain, defined as pain duration for at least three months with a mean score of 4 or higher on the Brief Pain Inventory (BPI) Pain Interference Scale
3. Pain severity of 4 or higher on a numerical rating scale (0-10) indicating "worst pain in the last week"
4. If using an antidepressant, the dose must be stable for the previous 2 months
5. Has received buprenorphine from the current primary care provider for at least the last month
6. Continuing buprenorphine with no plan to taper dose for the next 12 months
7. Score of ≥4 on Personal Health Questionnaire-9 instrument (at least "mild" depression severity)
8. Gives informed consent to participate in the study.

Exclusion Criteria:

1. Expected surgery in the next 3 months
2. Pain thought to be due to cancer, infection, or inflammatory arthritis
3. Greater than or equal to 10 days of cocaine/crack/methamphetamine use in the past month
4. Current (past month) mania or past year psychosis as determined via Structured Clinical Interview for DSM-5 (SCID) Module's A and B/C
5. Lifetime diagnosis of schizophrenia or other chronic psychotic condition as determined by the study PI
6. Planning to stop using buprenorphine in the next 6 months
7. Pregnancy or planned pregnancy in the next 6 months.
8. Greater than 8 homeless nights in the past month
9. Suicide ideation or behavior requiring immediate attention
10. Not able to provide informed consent
11. Not able to complete interviews in English
12. Unable to provide names and contact information for at least two verifiable locator persons who will know where to find them in the future.
13. Greater than or equal to 45 days without a phone in the past 3 months/no reliable access to phone
14. Headache/migraine as the only site of pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Stein, MD, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Stanley Street Treatment and Resources, Fall River, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stein MD, Bendiks S, Karzhevsky S, Pierce C, Dunn A, Majeski A, Herman DS, Weisberg RB. Study protocol for the Treating Opioid Patients' Pain and Sadness (TOPPS) study - A randomized control trial to lower depression and chronic pain interference, and increase care retention among persons receiving buprenorphine. Contemp Clin Trials. 2024 Aug;143:107608. doi: 10.1016/j.cct.2024.107608. Epub 2024 Jun 13. PMID 38878997
- [Derived] Haley DF, Stein MD, Bendiks S, Karzhevsky S, Pierce C, Dunn A, Herman DS, Anderson B, Weisberg RB. Associations of discomfort intolerance, discomfort avoidance, and cannabis and alcohol use among persons with chronic pain receiving prescription buprenorphine for opioid use disorder. Drug Alcohol Depend. 2024 Dec 1;265:112472. doi: 10.1016/j.drugalcdep.2024.112472. Epub 2024 Oct 24. PMID 39488941

RESULTS

PARTICIPANT FLOW:
Period: Allocation
Arm/Group | Treating Opioid Patients' Pain and Sadness (TOPPS) | Health Education (HE)
Started | 82 | 81
Completed | 82 | 81
Not Completed | 0 | 0
Period: Completed 3 Month Assessment
Arm/Group | Treating Opioid Patients' Pain and Sadness (TOPPS) | Health Education (HE)
Started | 82 | 81
Completed | 60 | 65
Not Completed | 22 | 16
Period: Completed 6 Month Assessment
Arm/Group | Treating Opioid Patients' Pain and Sadness (TOPPS) | Health Education (HE)
Started | 82 | 81
Completed | 66 | 64
Not Completed | 16 | 17
Period: Completed 9 Month Assessment
Arm/Group | Treating Opioid Patients' Pain and Sadness (TOPPS) | Health Education (HE)
Started | 82 | 81
Completed | 63 | 60
Not Completed | 19 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treating Opioid Patients' Pain and Sadness (TOPPS) | Health Education (HE) | Total
Number analyzed (Participants) | 82 | 81 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (10.8) | 43.7 (10.4) | 44.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 35 | 77
  Male | 40 | 46 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 67 | 74 | 141
  African American | 7 | 3 | 10
  Other | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 82 | 81 | 163
Pain Interference Based on the Brief Pain Inventory [Mean (Standard Deviation); unit: units on a scale] — Brief Pain Inventory- Interference Scale. Subscale of the Brief Pain Inventory. Measures pain's interference with physical and psychosocial functioning.
  Ranges from 0-10, with higher numbers indicating greater pain interference.
  units on a scale | 6.04 (1.57) | 6.02 (1.67) | 6.03 (1.61)
Pain Severity Based on the Brief Pain Inventory [Mean (Standard Deviation); unit: units on a scale] — Participants will indicate "average" pain in the last week. Scores range from 0-10 with higher scores indicating greater pain severity.
  units on a scale | 5.68 (1.66) | 5.68 (1.66) | 5.68 (1.66)
Patient Health Questionnaire- 9 Score [Mean (Standard Deviation); unit: units on a scale] — Objectifies degree of depression severity.
  Higher scores are indicative of higher levels of depressive symptoms.
  Scores range from 0-27.
  units on a scale | 12.33 (5.07) | 12.04 (4.96) | 12.18 (5.00)

OUTCOME MEASURES:

1. Primary Outcome: Pain Interference Based on the Brief Pain Inventory
Description: The Brief Pain Inventory Interference Scale (BPI-I) will be used to capture the domain of pain interference with physical and psychosocial functioning. The pain interference subscale includes 7 questions assessing the degree to which pain interferes with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life using a 0-to-10 numeric rating score. For interference items, 0 represents "does not interfere" and 10 indicates "interferes completely."
Time Frame: 3 Months
Population: These numbers represent those with non-missing data on the BPI-Interference subscale at 3 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treating Opioid Patients' Pain and Sadness (TOPPS) | Health Education (HE)
Number analyzed (Participants) | 59 | 64
units on a scale | 5.01 [4.54 to 5.47] | 4.67 [4.19 to 5.47]

2. Primary Outcome: Pain Severity Based on the Brief Pain Inventory
Description: Pain severity will be measured by the Visual Analogue Scale (VAS) presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." Participants will indicate "average" pain in the last week. Scores range between 0 and 10.
Time Frame: 3 Months
Population: These numbers represent those with non-missing data on the BPI at 3 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treating Opioid Patients' Pain and Sadness (TOPPS) | Health Education (HE)
Number analyzed (Participants) | 59 | 64
units on a scale | 5.17 [4.75 to 5.58] | 5.02 [4.65 to 5.39]

3. Primary Outcome: Depression Based on the Patient Health Questionnaire-9
Description: The Patient Health Questionnaire (PHQ-9) will be used to measure depression severity and suicidality. It is the major depressive disorder module of the full PHQ. Scores range from 0-27, with scores less than or equal to 4 suggesting minimal depression, scores from 5 to 9 indicating mild depression, 10 to 14 indicating moderately depression, 15 to 19 reflecting moderately severe depression, and scores greater than 20 indicating severe depression.
Time Frame: 3 Months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treating Opioid Patients' Pain and Sadness (TOPPS) | Health Education (HE)
Number analyzed (Participants) | 60 | 65
units on a scale | 10.91 [9.87 to 11.95] | 9.21 [8.13 to 10.30]

4. Secondary Outcome: Number of Participants Retained in Buprenorphine Treatment
Description: Using clinical records at the recruitment sites or participant self-report, we will assess whether participants were engaged in buprenorphine treatment at 12 months post study baseline
Time Frame: Month 12
Population: At month 12, data were available for 64 of the 82 participants in the TOPPS arm and 67 of the 81 participants in the HE arm for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treating Opioid Patients' Pain and Sadness (TOPPS) | Health Education (HE)
Number analyzed (Participants) | 64 | 67
Participants | 63 | 61

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of the 12-month study period.
Arm/Group | Treating Opioid Patients' Pain and Sadness (TOPPS) | Health Education (HE)
All-Cause Mortality (participants affected / at risk) | 1/82 | 1/81
Serious Adverse Events (participants affected / at risk) | 8/82 | 15/81
Other Adverse Events (participants affected / at risk) | 40/82 | 54/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treating Opioid Patients' Pain and Sadness (TOPPS) (N=82) | Health Education (HE) (N=81)
Hospitalization due to overdose (General disorders) | 1 (1) | 2 (2)
Hospitalization due to hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization- gallbladder removal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hospitalization due to sepsis (Infections and infestations) | 0 (0) | 2 (2)
Hospitalization due to lung infection (Infections and infestations) | 1 (1) | 0 (0)
Hospitalization due to myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Hospitalization due to pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Hospitalization- psychiatric (Psychiatric disorders) | 1 (1) | 3 (4)
Hospitalization due to severe back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hospitalization due to kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1)
Hospitalization- difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization due to fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization due to endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Hospitalization for flu symptoms (General disorders) | 1 (1) | 0 (0)
Hospitalization due to infection in foot (Infections and infestations) | 0 (0) | 1 (1)
Hospitalization due to pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Hospitalization due to lung inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization for substance use treatment (General disorders) | 1 (1) | 0 (0)
Hospitalization due to staph infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treating Opioid Patients' Pain and Sadness (TOPPS) (N=82) | Health Education (HE) (N=81)
Tooth abscess (Gastrointestinal disorders) | 1 (1) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 6 (8) | 5 (5)
Leg infection (Infections and infestations) | 1 (1) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Rib pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Withdrawal symptoms (General disorders) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Hand surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
ER visit- diabetes symptom management (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Tooth pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Influenza (General disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
RSV (Infections and infestations) | 1 (1) | 0 (0)
Respiratory infection (Infections and infestations) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Stomach virus (Gastrointestinal disorders) | 1 (2) | 2 (3)
Pneumonia (Infections and infestations) | 4 (5) | 2 (2)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (3)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood clot (Vascular disorders) | 2 (2) | 0 (0)
Fractured nose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sunburn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fractured wrist (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Motor vehicle accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Infection in arm (Infections and infestations) | 1 (1) | 0 (0)
Kidney stones (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchospasms (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Neck pain due to ablation (Infections and infestations) | 1 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Umbilical hernia (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fatigue (Nervous system disorders) | 1 (1) | 0 (0)
Hip dislocation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Toe infection (Infections and infestations) | 1 (1) | 0 (0)
Bleach in wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stroke symptoms (Nervous system disorders) | 1 (1) | 0 (0)
Eye disorder- other (Eye disorders) | 0 (0) | 2 (2)
COVID-19 infection (Infections and infestations) | 0 (0) | 2 (3)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Toe fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Difficulty breathing- asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Sinus infection (Infections and infestations) | 0 (0) | 3 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Facial wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 3 (3)
Strep throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Ear infection (Infections and infestations) | 0 (0) | 5 (5)
Injury from fight (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gallstone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Swollen lymph nodes (Infections and infestations) | 0 (0) | 1 (1)
Ankle sprain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Facial abscess/cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cyst on hand (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Finger wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Knee infection (Infections and infestations) | 0 (0) | 1 (1)
Forearm strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaginal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT03698669/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT03698669/ICF_000.pdf